CLINICAL TRIAL: NCT00047632
Title: Interferon Gamma-1b in Combination With Chemotherapy (Carboplatin/Paclitaxel) for First Line Therapy of Advanced Ovarian or Primary Peritoneal Carcinoma.
Brief Title: Safety and Efficacy of Interferon Gamma-1b Plus Chemotherapy for Ovarian and Peritoneal Cancer
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: futility
Sponsor: InterMune (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: GIOV-001
Record Dates: First submitted 2002-10-09; First posted 2002-10-11 (Estimated); Last update posted 2007-11-01 (Estimated); Status verified 2007-10

CONDITIONS: Ovarian Carcinoma; Peritoneal Carcinoma
Keywords: ovarian; carcinoma; peritoneal; cancer; ovary; interferon gamma
MeSH Terms: conditions — Ovarian Neoplasms; Carcinoma; Neoplasms | interventions — interferon gamma-1b

INTERVENTIONS:
Drug: Interferon gamma-1b — 100 mcg, SQ, 3x per week

SUMMARY:
The purposes of this study are to determine: 1) if treatment with interferon gamma-1b plus standard chemotherapy (carboplatin and paclitaxel) can increase the overall survival of patients with advanced ovarian or primary peritoneal carcinoma compared with chemotherapy alone; 2) how effective interferon gamma-1b plus standard chemotherapy is in preventing the progression or return of cancer; 3) the effects on quality of life; and 4) the safety of interferon gamma-1b combined with standard chemotherapy compared to chemotherapy alone.

DETAILED DESCRIPTION:
Approximately 800 patients will receive either chemotherapy alone or chemotherapy plus Interferon gamma-1b. Chemotherapy will be paclitaxel (175 mg/m2 over 3 hours) followed by carboplatin (AUC 6) every 3 weeks. Only those patients in the treatment arm will receive interferon doses. Interferon gamma-1b 100 mg will be administered subcutaneously 3 times per week (every other day; no more than 3 doses in a 7-day period) continuously while patients are treated with carboplatin / paclitaxel (including for the 3 weeks following the last dose of chemotherapy). A total of 6 cycles of chemotherapy will be given unless disease progression or liming toxicity occurs or patients refuse further treatment. Each patient will receive a total of 54 doses over a period of 18 weeks. Each patient's participation will be from 3-8 years in duration.

ELIGIBILITY:
Inclusion criteria:

* Histologically confirmed epithelial ovarian or primary peritoneal carcinoma, FIGO Stage III or IV disease. Patients with either optimal (<= 1 cm residual disease) or suboptimal residual disease following initial surgery are eligible. Unstained slides of the primary tumor, a primary tumor block, or cytological preparation must be available for review.
* Patients with the following histologic epithelial cell types are eligible: serous adenocarcinoma, endometrioid adenocarcinoma, mucinous adenocarcinoma, undifferentiated carcinoma, clear cell adenocarcinoma, mixed epithelial carcinoma, transitional cell carcinoma, malignant Brenner's Tumor, or adenocarcinoma N.O.S.
* <= 12 weeks after initial surgery with adequate recovery from surgery.
* Candidate for first-line chemotherapy
* Adequate bone marrow function (ANC >= 1,500/mL; platelets >= 100,000/mL; hemoglobin >= 10 gm/dL)
* Adequate hepatic function (AST, ALT, and alkaline phosphatase <= 2.5 x upper limit of normal; bilirubin <= 1.5 x upper limit of normal).
* Adequate renal function (creatinine <= 1.5 x upper limit of normal).
* Adequate neurologic function (sensory and motor neuropathy <= NCI CTC Grade 1).
* Negative urine pregnancy test in women of child-bearing potential (within 14 days of the initiation of the first chemotherapy cycle).
* Zubrod / ECOG / GOG performance score 0-2.
* Able to give informed consent.

Exclusion criteria:

* Epithelial ovarian tumors of low malignant potential (borderline carcinomas). If diagnosis is based on cytology alone [(e.g., fine needle aspiration (FNA)], slides must be available, and confounding carcinomas such as non-ovarian mucinous, colorectal, Fallopian tube, and other adenocarcinomas of non-ovarian origin must be ruled out.
* Prior therapy for ovarian or primary peritoneal carcinoma other than primary surgical debulking.
* Patients for whom therapy for ovarian or primary peritoneal carcinoma in addition to protocol therapy is planned.
* Prior biological response modifier (BRM) for any reason within the previous 5 years.
* Prior malignancy within the previous 5 years other than basal cell or squamous cell carcinomas or in situ carcinoma of the cervix. Patients who have had a malignancy > 5 years previously may be eligible for this trial if they have not received any anti-neoplastic treatment within the previous 5 years an dif they have been without any evidence of disease for the previous 5 years.
* Uncontrolled infection.
* Pregnant or nursing women are excluded. Women of child-bearing potential must agree to use a chemical or barrier contraceptive during the dosing portion of the study.
* Any illness or condition that in the opinion of the investigator may affect safety of treatment or evaluation of any of the study's endpoints.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 847 (Actual)
Dates: Start 2001-10; Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
Overall survival time assessed at end of study | 4 years

SECONDARY OUTCOMES:
Progression-free survival time assessed at interim analysis | 4 years
Treatment failure-free survival time assessed at end of study | 4 years
Quality of life assessed through 24 months after end of treatment | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: InterMune, Inc. 888-486-6411 — Medical Information
Locations (1):
- InterMune, Inc., Brisbane, California, United States